CLINICAL TRIAL: NCT01802515
Title: Atomoxetine Treatment for Opioid Maintained Cocaine Users
Brief Title: A Drug Treatment for Cocaine Users Who Are Also on Methadone Maintenance Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding stopped recruitment march 2014 with only 14 enrolled
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1206010407
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-07

CONDITIONS: Cocaine Dependence; Opiate Dependence
Keywords: addiction; cocaine; methadone; opiates; atomoxetine
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders; Behavior, Addictive | interventions — Atomoxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Atomoxetine, low dose (Active Comparator): 1 capsule containing 40mg of atomoxetine by mouth everyday for 8 weeks followed by 1 week of daily placebo capsules.
  Interventions: Drug: Atomoxetine, low dose
- Atomoxetine, high dose (Active Comparator): One capsule containing 80mg of atomoxetine by mouth everyday for 8 weeks, followed by 1 week of daily 40mg atomoxetine capsules
  Interventions: Drug: Atomoxetine, high dose
- Placebo (sugar pill) (Placebo Comparator): 1 placebo capsule by mouth everyday for 8 weeks of treatment invention followed by one week of placebo capsule during study medication taper.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine, low dose — The effects of 40mg low dose atomoxetine will be compared to placebo and to the 80mg atomoxetine high dose.
  Other Names: Strattera,; National Drug Codes - 00002-3229
  Arms: Atomoxetine, low dose
Drug: Atomoxetine, high dose — The effects of 80mg of high dose atomoxetine will be compared to placebo and to 40mg atomoxetine low dose.
  Other Names: Strattera, National Drug Codes - 00002-3250
  Arms: Atomoxetine, high dose
Drug: Placebo — The effects of placebo will be compared to the parallel groups of Atomoxetine high (80mg) dose and Atomoxetine low (40mg) dose.
  Other Names: sugar pill
  Arms: Placebo (sugar pill)

SUMMARY:
The main goal of this study is to evaluate the safety and tolerability of 40 or 80 mg atomoxetine as a treatment for cocaine dependence. The Phase I studies summarized above support the safety of atomoxetine in combination with stimulants. As the next step, the investigators will evaluate the safety and tolerability of atomoxetine in a small clinical trial with cocaine users. If atomoxetine is found to be promising in this study and sufficiently powered, double-blind, placebo-controlled studies will be proposed.

DETAILED DESCRIPTION:
This will be an approximately 13 to 14 week double-blind, placebo-controlled clinical trial testing the safety and feasibility of atomoxetine (40 or 80 mg/day) treatment, compared to placebo, in methadone-stabilized stimulant users. The study will have 3 phases: 1) a one to two week- methadone-induction phase; 2) an 8-week "treatment" phase; and 3) 1 week atomoxetine taper and about a 4-week methadone "taper and detoxification or transfer" phase. Subjects will be randomized to three treatment arms: 40 mg (n=15) atomoxetine, or 80 mg (n=15) atomoxetine, or placebo (n=15). During the methadone induction phase, subjects will be stabilized on methadone. During induction onto methadone, participants will be administered increasing doses of methadone starting at 30 mg daily, and this dose will be increased for stabilization of opiate withdrawal symptoms from 40 mg up to 140 mg depending on individual need. Based on the clinic schedule between 1 to 2 weeks after methadone treatment is initiated , atomoxetine treatment will be started at 40 mg/day. For those assigned to 80 mg of atomoxetine, the dose will be titrated up to 80 mg/day on the second week of treatment phase. At the end of the treatment-phase, subjects will undergo detoxification from methadone over a 4-week period based on an individual's needs, and they will concurrently be tapered off atomoxetine. All participants will receive a weekly one-hour of individual psychotherapy (Cognitive Behavioral Therapy) with experienced clinicians specifically trained to deliver the therapy, and who will receive ongoing supervision.

This study has been terminated as of march 2014 due to the lack of funding, only 14 were enrolled with 11 subject completers. (June 2016)

ELIGIBILITY:
Inclusion Criteria:

* • Men and women between 18 and 65 years old.

  * Current opioid dependence as evidenced by 1) documentation of prior treatment for opioid dependence or signs of withdrawal, 2) self-reported history of opioid dependence for 12 consecutive months and, 3) a positive urine toxicology screen for opiates.
  * Diagnosis of opioid dependence and cocaine dependence by Diagnostic and Statisical Manual (DSM-IV) -criteria as well as laboratory confirmation of recent cocaine use in the form of positive urine toxicology during the month prior to study entry.
  * For those who recently participated in a research study, at least 2 weeks of washout period before enrollment.
  * A history of cocaine use,( a minimum of 1/2 gram during the preceding 30 days).
  * Must be seeking treatment for opioid and cocaine use.
  * For women of childbearing age, a negative pregnancy test at screening with agreement to use adequate contraception to prevent pregnancy and monthly pregnancy tests.

Exclusion Criteria:

* • Serious medical illnesses including hypertension, tachycardia, bradycardia, or other arrhythmias and major cardiovascular, cerebrovascular, renal, endocrine, or hepatic disorders;

  * Serious psychiatric illness, history of psychosis, schizophrenia or bipolar type I disorder.
  * Current major depression. Subjects with current depressive symptoms not meeting criteria will be included in the study, with the exception of those endorsing suicidal and homicidal thoughts, will be excluded even if full criteria for major depression are not met.
  * Current diagnosis of alcohol or drug dependence other than opiates, cocaine, nicotine and cannabis.
  * Current use of over-the-counter or prescription psychoactive drugs (antidepressant, anxiolytics, antipsychotics, mood stabilizers, psychostimulants) or drugs that would be expected to have major interactions with drugs to be tested, e.g., benzodiazepines, codeine, percocet, and other opiate drugs that will interact with methadone.
  * Has not been treated with monoamine oxidase inhibitors within the last fourteen days.
  * Liver function tests (ALT or AST) greater than 3 times normal.
  * Known allergy or intolerance to atomoxetine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D,Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs Hospital, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female participants were recruited from the Greater New Haven area from September 2012 to January 2014 by word-of-mouth, flyers and from referrals from treatment centers in the local area. The study was conducted in an outpatient clinic of the West Haven VA Hospital.
Pre-assignment Details: After eligibility was determined, participants were randomized to placebo, 40 mg atomoxetine or 80 mg atomoxetine. The study consisted of 3 phases 1) a two-week methadone induction phase 2) an 8-week treatment phase and 3) a 4-week taper and detoxification or transfer phase.
Period: Overall Study
Arm/Group | Atomoxetine, Low Dose | Atomoxetine, High Dose | Placebo (Sugar Pill)
Started | 5 | 5 | 4
Completed | 2 | 5 | 4
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine, Low Dose | Atomoxetine, High Dose | Placebo (Sugar Pill) | Total
Number analyzed (Participants) | 5 | 5 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (8.0) | 47.6 (5.63) | 43.6 (0.95) | 42.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 7
  Male | 1 | 3 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Treatment Retention
Description: The number of participants completing all 8 weeks of treatment phase.
Time Frame: 8 weeks of treatment
Population: Descriptive statistics were calculated for all enrolled subjects. A full statistical analysis was not performed due to study termination.
Measure: Number; unit: participants
Arm/Group | Atomoxetine, Low Dose | Atomoxetine, High Dose | Placebo (Sugar Pill)
Number analyzed (Participants) | 5 | 5 | 4
participants | 2 | 5 | 4

2. Secondary Outcome: Change Score in the Center for Epidemiological Studies-Depression (CES-D) Scale
Description: Center for Epidemiological Studies-Depression. The CES-D is a 20-item self-report measure of depressive symptoms. Each of the 20 items can yield a score from 0 to 3 for a maximum total CES-D score of 60. Larger values represent more severe symptoms. It is a validated instrument with a score of 16 or more indicating clinically significant depression. The CES-D change score was computed as (total baseline CES-D score - total CES-D score at end of study).
Time Frame: 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine, Low Dose | Atomoxetine, High Dose | Placebo (Sugar Pill)
Number analyzed (Participants) | 2 | 5 | 4
units on a scale | -2.2 (5.2) | -2.2 (9.1) | -3.3 (11.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected once per week on all enrolled subjects for the 8 weeks of the treatment phase.
Description: The assessment of adverse events utilized the Brief Symptom Inventory (BSI), an instrument that consists of 77 items.
Arm/Group | Atomoxetine, Low Dose | Atomoxetine, High Dose | Placebo (Sugar Pill)
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 2/5 | 4/5 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine, Low Dose (N=5) | Atomoxetine, High Dose (N=5) | Placebo (Sugar Pill) (N=4)
insomnia (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
cramps (Reproductive system and breast disorders) | 1 (8) | 0 (0) | 0 (0)
dry mouth (Nervous system disorders) | 1 (4) | 2 (10) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (8) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (7) | 0 (0)
chills (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
heartburn (Gastrointestinal disorders) | 0 (0) | 1 (8) | 0 (0)
yawning (Nervous system disorders) | 0 (0) | 1 (8) | 0 (0)
agitation (Nervous system disorders) | 1 (3) | 3 (6) | 0 (0)
depression (Nervous system disorders) | 0 (0) | 3 (9) | 1 (5)
tiredness (Nervous system disorders) | 0 (0) | 3 (6) | 1 (4)
anxiety (Nervous system disorders) | 1 (1) | 2 (5) | 0 (0)
decreased libido (Nervous system disorders) | 0 (0) | 1 (8) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (3) | 2 (4) | 0 (0)
increased perspiration (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
decreased appetite (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0)
nightmares (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
numbness (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0)
decreased concentration (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
drowsiness (Nervous system disorders) | 0 (0) | 2 (10) | 1 (2)
hallucinations (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
tingling (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated after 14 subjects enrolled. 11 completers. 3 subjects dropped out in treatment week 7. There were no serious adverse events. Only descriptive statistics were computed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No